CLINICAL TRIAL: NCT01044381
Title: A Phase 1/2a, Open-Label Study Evaluating the Pharmacokinetics, Safety and Tolerability of Luliconazole Solution, 10% in Subjects With Moderate to Severe Distal Subungual Onychomycosis
Brief Title: Open-Label Pharmacokinetics (PK)/Safety Study of Luliconazole Solution, 10% in Distal Subungual Onychomycosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Topica Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0901-S
Record Dates: First submitted 2010-01-04; First posted 2010-01-07 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Onychomycosis
Keywords: Toenail; Fungal Infections; DSO
MeSH Terms: conditions — Onychomycosis; Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Luliconazole Solution, 10% (Experimental)
  Interventions: Drug: Luliconazole Solution, 10%

INTERVENTIONS:
Drug: Luliconazole Solution, 10% — 28 days of daily application

SUMMARY:
To determine the safety, tolerability, systemic exposure and pharmacokinetics of luliconazole after repeat daily topical application of Luliconazole Solution, 10% in a maximal use setting in adults with distal subungual onychomycosis of the toenails.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Distal Subungual Onychomycosis(DSO)on both great toenails with >=50%involvement of at least 1 great toenail
* At least 4 additional toenails with DSO
* Positive KOH and culture
* Normal renal and hepatic function

Exclusion Criteria:

* Subjects with hypersensitivity to imidazole compounds or any other ingredient
* Subjects unwilling to refrain from use of nail cosmetics until end of study
* Subjects with symptomatic tinea pedis
* Subjects with any history of cardiac disease of cardiac rhythm abnormalities
* Female subjects who are pregnant, nursing, or planning a pregnancy
* Subjects who have not undergone the specified washout period(s) for the following or requiring the concurrent use of: topical antifungal within 4 weeks; topical anti-inflammatory, corticosteroids, topical immunomodulators within 2 weeks; systemic corticosteroids within 2 weeks; systemic immunomodulators within 4 weeks.
* Subjects receiving systemic antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophytes within the previous 12 weeks or 5 half-lives of the drug, whichever is longer
* Subjects receiving any other treatment/therapy for the onychomycosis not previously mentioned (e.g., laser treatment) within 4 weeks
* Subjects with a history of significant internal disease or with a life threatening condition within the last 6 months
* Subjects with anatomic abnormalities of the toe(s) and or toenails
* Subject who have donated or lost a large volume of blood (~500 mL or more, during the previous 6 weeks
* Subjects with a recent history of or currently known to abuse drugs or alcohol
* Subjects currently participating in another investigational medication or device study or have participated in a clinical trial within 30 days or five half-lives of the test medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
PK parameters (AUC, Cmax, Tmax, t1/2) will be measured at days 1 (Baseline), 9, 15 and 29. Safety assessments include monitoring of adverse events, local site tolerability, ECG monitoring, and changes in laboratory values and vital signs. | March 2011

SECONDARY OUTCOMES:
Evaluation of linear toenail growth. | March 2011

CONTACTS AND LOCATIONS:
Overall Officials: Terry M Jones, M.D., Principal Investigator — J&S Studies
Locations (1):
- J&S Studies, College Station, Texas, United States